CLINICAL TRIAL: NCT06040060
Title: Effects of Ketamine 0.5 Mg/Kgbw Administration as Preemptive Analgesia on Analgesia Duration and the Need for Fentanyl Following Hysterectomy Surgery
Brief Title: Ketamine Effects as Preemptive Analgesia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AN-202309.02
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Pain, Postoperative
Keywords: Ketamine; Preemptive Analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preemptive Ketamine (Active Comparator): Preemptive administration of Ketamine 0.5 mg/kgBB intravenously, given 10 minutes prior to incision
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Placebo administration of 10 mL NaCl 0,9% intravenously, given 10 minutes prior to incision
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine — The intervention was prepared by the research team (anesthesia resident) in the form of ketamine which had been diluted to a dosage of 10 mg/cc, taken according to the required dose based on actual body weight then diluted with 0.9% NaCl to 10 cc. Then the two solutions were given to researchers without knowing the contents of the drugs that had been prepared by the resident who assisted in this research.
  Arms: Preemptive Ketamine
Other: Placebo — While the 0.9% NaCl solution was used as placebo was prepared in a 10 cc syringe
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled trial is to compare the effect of preemptive ketamine administration to placebo administration in patients underwent hysterectomy surgery. The main questions it aims to answer are:

1. To determine the effect of ketamine at a dose of 0.5 mg/kgBW as preemptive analgesia on the duration of analgesia after hysterectomy surgery
2. To determine the effect of ketamine at a dose of 0.5 mg/kgBW as preemptive analgesia on the need for fentanyl after hysterectomy surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-50 years.
2. ASA I and II physical status (American Society of Anesthesiologists).

Exclusion Criteria:

1. The patient is not willing to be included as a research subject
2. The patient takes anti-pain medication before surgery
3. History of allergies to the drugs to be used
4. History of chronic pain

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women only
Enrollment: 40 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | 24 hours post operative
  Time interval from completion of hysterectomy until additional analgesic is needed, namely fentanyl 25 µg via PCA
Total need for post-operative analgesic rescue | 24 hours post operative
  The total amount of rescue analgetic required by research subjects, during the 24 hours after surgery, was given via PCA

CONTACTS AND LOCATIONS:
Overall Officials: Iwan Fuadi, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Ardi Zulfariansyah, MD, Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Jacklin E Mokoginta, MD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Universitas Padjadjaran, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No